CLINICAL TRIAL: NCT02764164
Title: Transcranial Direct Current Stimulation for Auditory Hallucinations in Early Onset Schizophrenia
Brief Title: Transcranial Direct Current Stimulation (TDCS) for Auditory Hallucinations in Early Onset Schizophrenia (EOS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-6134
Record Dates: First submitted 2015-08-03; First posted 2016-05-06 (Estimated); Results first posted 2020-10-20 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2016-09

CONDITIONS: Schizophrenia
Keywords: TDCS
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention Active tDCS (Experimental): Affected subjects receiving up to 2 milliamps (mA) active tDCS, open label
  Interventions: Device: Intervention Active tDCS

INTERVENTIONS:
Device: Intervention Active tDCS — Transcranial direct current stimulation (tDCS) is a form of neurostimulation which uses constant, low current delivered directly to the brain area of interest via small electrodes. Placed over the temporoparietal junction to suppress auditory hallucinations.
  Other Names: tdcs

SUMMARY:
Youths diagnosed with early onset schizophrenia will demonstrate amelioration of auditory hallucinations after one week of twice daily treatment with transcranial direct current stimulation (tDCS).

DETAILED DESCRIPTION:
Background: Early onset schizophrenia (EOS) involves positives symptoms such as psychotic behaviors, as well as negative symptoms such as disruptions to normal emotions and behaviors. Antipsychotics are the primary method of treatment in pediatric populations, but can produce unpleasant or dangerous side effects. Medication response is highly variable. Recent evidence demonstrates transcranial Direct Current Stimulation (tDCS) relieving auditory hallucinations (AH) associated with schizophrenia in adults, and to a lesser degree negative and cognitive symptomology. Such studies provide important scientific and technical knowledge that may be applied to pediatric populations.

Hypothesis: 1. Primary: Youths with EOS will demonstrate amelioration of AH after administration of tDCS. 2. TDCS will be well-tolerated in pediatric populations with minimal adverse side effects.

ELIGIBILITY:
Inclusion Criteria:

* Structured Clinical Interview for Diagnostic and Statistical Manual (DSM) Disorders (SCID) primary diagnosis of DSM-IV (Diagnostic and Statistical Manual of Mental Disorders-Version IV) schizophrenia or schizoaffective disorder
* Ages 8 to 25 years-old
* Persistent auditory hallucinations
* Full Scale intelligent quotient (IQ) greater than 60.
* Stable antipsychotic medication for > 4 weeks
* If female and not infertile patient must agree to use one of the following forms of contraception for the duration of study participation: systemic hormonal treatment or an interuterine device (IUD).
* Legal guardian has provided written informed consent and the subject has provided written informed assent when able. Expectation that a majority of subjects will be able to assent but the potential for the younger children and/or those that are of borderline intellectual functioning will not be able to assent.

Exclusion Criteria:

* History of alcohol, substance dependence or abuse in the past 90 days
* Open skin wounds that would preclude use of TDCS electrodes
* If female, pregnancy or breast feeding, as determined during eligibility pre-screen call
* Subjects exhibiting significant ongoing severe disruptive, aggressive, self-injurious, or sexually inappropriate behavior will not be eligible for enrollment.
* Presence of any medical condition that would make treatment with tDCS less safe. This includes any implanted metal device or any cardiac pacemaker. Subjects with a history of a seizure disorder are permitted if the subject has been seizure free for 6 months and is currently treated with an anticonvulsant that has been stable for 4 weeks.
* Presence of any other condition that would make the participants unable to comply with the requirements of the study for any reason. This may include an appreciable hearing or visual impairment.

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Pedapati, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brunelin J, Mondino M, Gassab L, Haesebaert F, Gaha L, Suaud-Chagny MF, Saoud M, Mechri A, Poulet E. Examining transcranial direct-current stimulation (tDCS) as a treatment for hallucinations in schizophrenia. Am J Psychiatry. 2012 Jul;169(7):719-24. doi: 10.1176/appi.ajp.2012.11071091. PMID 22581236

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Active tDCS
Started | 1
Completed | 1 (Duration flexible up to 12mo, ended early (funding), 2 week time point achieved)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Active tDCS
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Severity of Auditory Hallucinations Measured by Auditory Hallucinations Rating Scale
Description: The primary efficacy assessment is the mean change from baseline to the last observed post-baseline visit in total score on the Auditory Hallucination Rating Scale (AHRS). Minimum score is 2, maximum score is 41, higher score indicates more severe symptoms.
Time Frame: Baseline to last observation: at baseline, following 5 days of TDCS, pre-specified every 3 months for up to 12 months, 2 week time point achieved
Population: Entire time period was not achieved; participant was only followed for 2 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Active tDCS
Number analyzed (Participants) | 1
score on a scale
  Baseline | 31 (0)
  Same day post TDCS | 20 (0)
  2 weeks post baseline | 17 (0)
  3 months post baseline: number analyzed (Participants) | 0
  6 months post baseline: number analyzed (Participants) | 0
  9 months post baseline: number analyzed (Participants) | 0
  12 months post baseline: number analyzed (Participants) | 0

2. Secondary Outcome: Change in Schizophrenia Symptom Type as Measured by the Positive and Negative Syndrome Scale (PANSS)
Description: The primary secondary outcome measure will be the change in severity of other symptoms of schizophrenia, assessed using the Positive and Negative Syndrome Scale (PANSS) from baseline to last observation, expected average of every 3 months. The PANSS can be computed as a dimensional scale including positive, negative, depression, disorganization, and grandiosity/excitement. Both the positive and negative scales have minimum scores of 7 and maximum scores of 49. The general scale has a minimum score of 16 and a maximum score of 112. Total score minimum is 30 and total score maximum is 210. Higher scores indicate more severe symptoms.
Time Frame: Baseline to last observation: at baseline, following 5 days of TDCS, and pre-specified 1, 3, and 6 months, expected average of 3 months for us to 12 months, post-TDCS timepoint achieved
Population: Entire time period was not achieved; participant was only followed for 2 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Active tDCS
Number analyzed (Participants) | 1
units on a scale
  Baseline | 87 (0)
  Same day post TDCS | 78 (0)
  1 month post baseline: number analyzed (Participants) | 0
  3 months post baseline: number analyzed (Participants) | 0
  6 months post baseline: number analyzed (Participants) | 0
  9 months post baseline: number analyzed (Participants) | 0
  12 months post baseline: number analyzed (Participants) | 0

3. Secondary Outcome: Change in Disorder Severity as Measured by Clinical Global Impressions Severity Scales (CGI-S)
Description: Mean change from baseline to the last observed post-baseline visit Clinical Global Impression (CGI-S) severity scales. The minimum score on the CGI-S is 1 and the maximum score is 7. A higher score indicates more severe illness.
Time Frame: Baseline to last observation: at baseline, following 5 days of TDCS, pre-specified at 1, 3, and 6 months, expected average of 3 months for up to 12 months, post-TDCS time point achieved
Population: Entire time period was not achieved; participant was only followed for 2 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Active tDCS
Number analyzed (Participants) | 1
score on a scale
  Baseline | 6 (0)
  Same day post TDCS | 6
  1 month post baseline: number analyzed (Participants) | 0
  3 months post baseline: number analyzed (Participants) | 0
  6 months post baseline: number analyzed (Participants) | 0
  9 months post baseline: number analyzed (Participants) | 0
  12 months post baseline: number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Intervention Active tDCS
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes